CLINICAL TRIAL: NCT05094284
Title: BioFreedom Ultra Stent in Hong Kong All Comers Registry
Brief Title: BioFreedom Ultra Registry
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Other Study IDs: 2021.459
Record Dates: First submitted 2021-10-17; First posted 2021-10-26 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Disease
Keywords: BioFreedom Ultra; Drug-eluting stent; percautaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BioFreedom Ultra — this is a registry only

SUMMARY:
Over the past three decades, coronary stent struts have been made progressively thinner. Thin strut drug-eluting stents (DES) performed better than their thicker counterparts in a recent study. Thinner struts discourage abnormal coronary flow after implantation and associated with greater flexibility, deliverability and better clinical outcomes. Lower strut thickness may be particularly advantageous in small target vessels because thicker struts and smaller minimum in-stent lumen diameter are independent predictors of in-stent restenosis.

BioFreedom Ultra is a thin strut (84μm), cobalt-chromium, carrier-free drug-coated stent with Biolimus A9 drug. The BioFreedom Ultra stent is intended for percutaneous coronary intervention (PCI) for high-bleeding-risk (HBR) patients treated with 1-month dual antiplatelet therapy. BioFreedom Ultra received CE mark in October 2020 supported by the LEADERS FREE III trial which enrolled 400 HBR patients using the same inclusion criteria as the LEADERS FREE randomized trial. LEADERS FREE III is a single-arm trial, with all patients treated using the BioFreedom Ultra stent. The data was compared to the BioFreedom stainless steel drug-coated stent (DCS-StS) and bare-metal stent (BMS) groups from LEADERS FREE. The primary safety endpoint of the trial was a composite of cardiac death, myocardial infarction, or definite/probable stent thrombosis. The primary efficacy endpoint was clinically driven target lesion revascularization. The study found that the BioFreedom Ultra was non-inferior to the DCS-StS for safety and superior to the BMS for efficacy. Definite or probable stent thrombosis at 1 year in this HBR population was only 1%. Recently, the Biofreedom QCA randomized trial compared the Biofreedom Ultra with the stainless steel version (DCS-StS) in an all-comer population. In this prospective, single-blind non-inferiority randomized (1:1) trial, BioFreedom Ultra was non-inferiority for late lumen loss at 9 months in comparison with DCS-StS.

ELIGIBILITY:
Inclusion Criteria:

This is an "all comers" registry and patient who will be enrolled have to meet following criteria:

* Patient must be at least 18 years of age
* Patient must have indication to percutaneous coronary intervention including:

  * Stable angina or evidence of myocardial ischemia with stress echocardiography/ myocardial SPECT/exercise test, or
  * Unstable angina / non ST-elevation myocardial infarction, OR
  * ST-elevation myocardial infarction with de novo culprit lesion.
* Presence of one or more coronary artery stenosis >50% with reference diameter 2.0-6.0mm which can be covered by one or multiple stents

Exclusion Criteria:

* Known intolerance to any of the device components
* Inability to provide written informed consent
* Participating in other trial before reaching primary endpoint
* Planned surgery within 1 month of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Being an observational registry aiming to quantify effect estimates without direct comparisons to other devices, we used confidence interval profiling for sample size justification. Assuming an 8.43% MACE rate at 1 year [5], 95% confidence intervals computed with the adjusted Wald method would be 5.4% to 11.5% for a 300 patient sample. Given that the registry aims to reflect real-world patients and practice, 300 patients will be enrolled in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
MACE events | 12 months post index procedure
  12-months cumulative hierarchical incidence of major adverse cardiac events (MACE) defined as: cardiac death, non-fatal myocardial infarction (MI) and clinically indicated target vessel revascularization (TVR). In order to minimize bias in assessing MACE outcomes, these events will be adjudicated by an independent observer.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sabate M, Okkels Jensen L, Tilsted HH, Moreno R, Garcia Del Blanco B, Macaya C, Perez de Prado A, Cequier A, Perez-Fuentes P, Schutte D, Costa RA, Stoll HP, Flensted Lassen J. Thin- versus thick-strut polymer-free biolimus-eluting stents: the BioFreedom QCA randomised trial. EuroIntervention. 2021 Jun 25;17(3):233-239. doi: 10.4244/EIJ-D-20-01162. PMID 33433389
- [Result] Buiten RA, Ploumen EH, Zocca P, Doggen CJM, van der Heijden LC, Kok MM, Danse PW, Schotborgh CE, Scholte M, de Man FHAF, Linssen GCM, von Birgelen C. Outcomes in Patients Treated With Thin-Strut, Very Thin-Strut, or Ultrathin-Strut Drug-Eluting Stents in Small Coronary Vessels: A Prespecified Analysis of the Randomized BIO-RESORT Trial. JAMA Cardiol. 2019 Jul 1;4(7):659-669. doi: 10.1001/jamacardio.2019.1776. PMID 31111862
- [Result] Urban P, Meredith IT, Abizaid A, Pocock SJ, Carrie D, Naber C, Lipiecki J, Richardt G, Iniguez A, Brunel P, Valdes-Chavarri M, Garot P, Talwar S, Berland J, Abdellaoui M, Eberli F, Oldroyd K, Zambahari R, Gregson J, Greene S, Stoll HP, Morice MC; LEADERS FREE Investigators. Polymer-free Drug-Coated Coronary Stents in Patients at High Bleeding Risk. N Engl J Med. 2015 Nov 19;373(21):2038-47. doi: 10.1056/NEJMoa1503943. Epub 2015 Oct 14. PMID 26466021
- [Result] Garot P, Morice MC, Tresukosol D, Pocock SJ, Meredith IT, Abizaid A, Carrie D, Naber C, Iniguez A, Talwar S, Menown IBA, Christiansen EH, Gregson J, Copt S, Hovasse T, Lurz P, Maillard L, Krackhardt F, Ong P, Byrne J, Redwood S, Windhovel U, Greene S, Stoll HP, Urban P; LEADERS FREE Investigators. 2-Year Outcomes of High Bleeding Risk Patients After Polymer-Free Drug-Coated Stents. J Am Coll Cardiol. 2017 Jan 17;69(2):162-171. doi: 10.1016/j.jacc.2016.10.009. Epub 2016 Oct 30. PMID 27806919